CLINICAL TRIAL: NCT03035136
Title: Retrospective Study on Epidemiology of Colorectal Lesions
Status: Completed | Type: Observational
Sponsor: Lyell McEwin Hospital (Other Government)
Responsible Party: Principal Investigator, Leonardo Zorron Cheng Tao Pu, Principal Investigator, Lyell McEwin Hospital
Other Study IDs: SSA/17/NALHN/3
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: ColoRectal Cancer; Colonic Polyp; Colonic Neoplasms
Keywords: polyps
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps; Colonic Neoplasms; Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with colorectal lesions: Patients with a full colonoscopy that showed either a cancer or a polyp.
- Patients without colorectal lesions: Patients with a full colonoscopy that showed no polyps.

SUMMARY:
Retrospective analysis on colonoscopies in the endoscopy unit of the Lyell McEwin Hospital.

DETAILED DESCRIPTION:
Colonoscopy reports will be manually searched by the investigator to evaluate epidemiology on colorectal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopies performed in Lyell McEwin Hospital between 2010-2016

Exclusion Criteria:

* Sigmoidoscopies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All colonoscopies performed in Lyell McEwin Hospital between 2010 and 2016.
Sampling Method: Non-Probability Sample
Enrollment: 2658 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | Day 1
  Percentage of screening patients with at least one adenomatous lesion found - to be compared between Gastroenterologists and Surgeons and based on scheduling of the procedure

SECONDARY OUTCOMES:
SSA/P detection rate | Day 1
  Percentage of screening patients with at least one SSA/P found - to be compared between Gastroenterologists and Surgeons and based on scheduling of the procedure
Polyp detection rate | Day 1
  Percentage of screening patients with at least one polyp found - to be compared between Gastroenterologists and Surgeons and based on scheduling of the procedure

IPD SHARING:
Plan to Share IPD: No